CLINICAL TRIAL: NCT04923061
Title: The Effect of Acupressure on Sleep Quality and Fatigue in Nurses Working in Internal Clinics During the COVID-19 Pandemic Process: A Randomized Controlled Study
Brief Title: The Effect of Acupressure on the Sleep Quality and Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Esra Cavusoglu, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MersinUniversityNursing
Record Dates: First submitted 2021-06-05; First posted 2021-06-11 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Sleep; Fatigue
Keywords: Acupressure; Sham acupressure; Nurse; Sleep quality; Fatigue
MeSH Terms: conditions — Fatigue; Sleep Initiation and Maintenance Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: As a result of the draw, group A was determined as acupressure and group B as sham acupressure group. Information showing that the nurses included in the research sample were assigned to groups A and B according to the randomization table will be placed in an opaque envelope. This envelope will be kept by the coordinator researcher (MG) and when the researcher with acupressure practice certificate (EC) goes to the nurse for the application, fills out the "Informed Consent Form" and opens the envelope to find out which group the nurse is in. Since all nurses included in the study will be taught to apply pressure to the pressure point, the participants will be blinded as the nurses do not know whether acupressure or sham acupressure is applied. The researcher (EC) cannot be blinded due to the nature of the research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): The experimental group will apply acupressure to themselves three times a week for a total of 12 sessions for four weeks.
  Interventions: Other: Acupressure
- Sham acupressure group (Sham Comparator): The sham group will apply acupressure to themselves three times a week for a total of 12 sessions for four weeks.
  Interventions: Other: Sham acupressure group

INTERVENTIONS:
Other: Acupressure — In the acupressure group, heart meridian 7th point (HT7), large intestine meridian 4th point, stomach meridian 36th point (ST36) and spleen meridian 6th point (SP6) will be applied. Tissue sensitivity will be reduced by heating and rubbing for about 20 seconds without direct pressure on the acupressure points, and the points will be ready for acupressure application. Subsequently, consecutive (breathing rhythm) compressions will be applied to the acupressure points determined by the researcher, without raising the finger, taking into account the pain threshold of the individual who is applied with the thumb, with 10 seconds of pressure for two seconds of relief Since the symmetry of the selected four different points will also be applied to the other extremity, a total of 16 minutes of compression will be applied to each point, provided that it is two minutes. Each nurse's session will be approximately 20 minutes, depending on the preparation and compression time on each point.
  Arms: Acupressure group
Other: Sham acupressure group — In the sham group, acupressure will be applied on the bone region where the meridians do not pass, approximately 1-1.5 cm away from the HT7, LI4, ST36, SP6 points. The application process will continue in the same way with acupressure group and the pressure intensity will be less.
  Arms: Sham acupressure group

SUMMARY:
This research aims to determine the effect of acupressure applied to nurses actively working in internal clinics on sleep quality and fatigue during the COVID-19 pandemic process. This research hypothesizes that acupressure improves sleep quality and reduces fatigue.

DETAILED DESCRIPTION:
In this study, 68 nurses working in internal clinics were randomly assigned to acupressure and placebo (sham) acupressure groups. In the acupressure group (n=34), the heart meridian 7th point (HT7), large intestine meridian 4th point (LI4), stomach meridian 36th point (ST36) and spleen meridian 6th point (SP6) will be applied to a total of four points. Depending on the preparation and compression time on each point, the session duration of each nurse will be 20 minutes on average. In the sham group (n=34), pressure will be made approximately 1-1.5 cm away from the HT7, LI4, ST36, SP6 points. In the Sham group, the acupressure application time will take 20 minutes on average. Reminder text messages (SMS) will be sent before the application on the days when the nurses will practice, so that they continue to do the application regularly. At the end of the application, after the data collection process is completed, the sham group will be taught the correct acupressure points. Nurses will apply acupressure three times a week for a total of 12 sessions for four weeks. The primary outcome of the research is the effect of acupressure on the sleep quality of nurses. The secondary outcome of the study is to determine the effect of acupressure on fatigue. The outcomes will be collected before and four weeks after the acupressure and sham acupressure administration.

ELIGIBILITY:
Inclusion Criteria:

Nurses who care for COVID 19 patients during the pandemic process

Nurses working in internal clinics during the data collection process

Those who have recovered from COVID 19

Those who agreed to participate in the study

No deformity or lesions in the areas where acupressure will be applied

No acupressure experience

No sleep disorder diagnosis and no medical treatment

Not diagnosed with anxiety disorder and not receiving medical treatment

Not diagnosed with depression and not receiving medical treatment

Coffee, cigarette and alcohol free

No mental disorder

Night shift workers

Those who can understand and speak Turkish

Those who signed the Informed Consent Form

Exclusion Criteria:

Nurses who did not work in internal clinics during the data collection process

Nurses who do not care for COVID 19 patients during the pandemic process

Those with active COVID 19

Those who do not agree to participate in the study

Those who have any deformity or lesion in the areas where acupressure will be applied

Experiences of acupressure

Heart and kidney failure, severe anemia, immunodeficiency problem

Pregnant

Diagnosed with sleep disorder and receiving treatment

Anxiety disorder and treatment

Depression diagnosed and treated

Coffee, cigarette and alcohol addiction

Having mental illness

Fixed day shift workers

Those who can not understand and speak Turkish

Those who did not sign the Informed Consent Form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Sleep quality evaluated using the Pittsburgh Quality Sleep Index | Change from before implementation and 4th week of practice.
  The total scale score is in the range of 0 (minimum) -21 (maximum), and the high total Pittsburgh Quality Sleep Index (PSQI) score indicates that sleep quality is low. A total PSQI score between 0-4 indicates good sleep quality, while between 5-21 shows that sleep quality is low.

SECONDARY OUTCOMES:
Fatigue evaluated using the Fatigue Severity Scale | Change from before implementation and 4th week of practice
  It is a Likert-type scale consisting of a total of nine items, each item being evaluated between 1 and 7 (1=I totally disagree, 7=I totally agree). The fatigue score is obtained by dividing the total score obtained from the scale by the number of scale items. The score that can be obtained from the scale varies between 9 and 63. A high score indicates an increased level of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Gun, Doctorate, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No